CLINICAL TRIAL: NCT06257862
Title: Translation, Cross-cultural Validity and Reliability of a Danish Version of the Anterior Knee Pain Scale (Kujala-DK)
Brief Title: Translation, Cross-cultural Validity and Reliability of a Danish Version of the Anterior Knee Pain Scale
Acronym: Kujala-DK
Status: Active, not recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Lind, Professor, PhD, MD, Aarhus University Hospital
Other Study IDs: Questionnaire KUJALA-DK
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Patella Subluxation; Patellofemoral Pain Syndrome
Keywords: MPFL; KUJALA; PAIN; Questionnaire; TRANSLATION
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Anterior Knee Pain Scale (Kujala) is a questionnaire designed to assess adults with patellofemoral disorders and is widely used in both anterior knee pain and patellar dislocation patients.The questionnaire is a patient-reported outcome measure (PROM), that was developed in 1993 and has been translated and validated into most major languages (e.g. French, Italian, Chinese, German, and Spanish) and has gained wide international acceptance. In a recent systematic review, the Kujala was among the eight most commonly used PROMS for patients with patellofemoral pain. In addition, the Kujala was used in almost 80% of studies of patellofemoral instability/dislocation.

The Kujala has been widely used in Denmark during the last 15 years, but surprisingly it has not been translated and validated in Danish according to international guidelines. The translation of the Kujala into Danish will stimulate to more valid and precise results of the Kujala questionnaire in both patients with anterior knee pain and patients with patellar dislocation

The aim of this study is to cross-cultural translate and adapt the Kujala into a Danish Kujala-DK. Secondarily to determine validity and reliability of the Kujala-DK in two consecutive Danish populations of patients with either anterior knee pain or patellar dislocation.

ELIGIBILITY:
Inclusion Criteria:

* Danish speaking
* MPFL-reconstructed

Exclusion Criteria:

-

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: MPFL-reconstructed patients.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Kujala (Anterior Knee Pain Scale) | Baseline, after 6-8 days
  Patient reported outcome score. (0-100 (0 = Worst, 100 = Best)
Victorian Institute of Sports Assessment - Patella questionnaire (VISA-P) | Baseline
  Patient reported outcome score. (0-100 (0 = Worst, 100 = Best)
International knee documentation committee (IKDC) | Baseline
  Patient reported outcome score. (0-100 (0 = Worst, 100 = Best)
Banff patella instability instrument (BPII 2.0) | Baseline
  Patient reported outcome score. (0-100 (0 = Worst, 100 = Best)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Sports Trauma, Palle Juul-Jensens Boulevard 99, Aarhus N, Denmark